CLINICAL TRIAL: NCT03675854
Title: Defining the Optimal Duration of Treatment for "Low-Risk" Peritoneal Dialysis-Related Peritonitis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: New data from another study show that a positive result is unlikely.
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheuk-Chun SZETO, Professor, Department of Medicine & Therapeutics, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CREC-2018.245-T
Record Dates: First submitted 2018-09-17; First posted 2018-09-18 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Peritoneal Dialysis-associated Peritonitis
Keywords: end stage renal disease; infection; antibiotic
MeSH Terms: conditions — Kidney Failure, Chronic; Infections | interventions — Cefazolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extended Group (Experimental): 3 weeks of antibiotics
  Interventions: Drug: Cefazolin
- Conventional Group (Active Comparator): 2 weeks of antibiotics
  Interventions: Drug: Cefazolin

INTERVENTIONS:
Drug: Cefazolin — 3 weeks

SUMMARY:
Background According to the International Society for Peritoneal Dialysis (ISPD) recommendations, "low-risk" peritoneal dialysis (PD)- related peritonitis caused by coagulase-negative staphylococcal species, Streptococcal species, or negative bacterial culture should receive antibiotics for 2 weeks. However, relapsing, recurrent, or repeated episodes are common.

Objectives To compare the incidence of relapsing, recurrent, and repeat peritonitis with a 3-week course, as compared to the conventional 2-week course, antibiotic for PD-related peritonitis. Hypothesis Treatment of low-risk PD-related peritonitis for 3 weeks reduces the incidence of relapsing, recurrent, and repeat peritonitis. Design and subjects Randomized control trial of 310 episodes of "low-risk" PD-related peritonitis.

Study instruments and interventions Patients will be randomized to receive treatment of the effective antibiotic according to the ISPD recommendations for 2 weeks (Conventional Group) or 3 weeks (Extended Group). All patients will be followed for 6 months after completion of treatment. Main outcome measures Complete cure of the peritonitis episode, defined as survival for 6 months without relapsing, recurrent, or repeat peritonitis episodes. Data analysis Data will be analyzed by both intention-to-treat and per protocol approach. The incidences of complete cure, relapsing, recurrent, and repeated peritonitis episodes will be compared. Expected results Based on our pilot study, we expect to find a significantly lower rate of relapsing, recurrent, and repeated peritonitis episodes in the Extended Group. By proving that "low-risk" peritonitis episodes require 3-week course of antibiotic therapy, our result will change the current recommendation and make treatment for 3 weeks course the standard of care.

DETAILED DESCRIPTION:
Background According to the International Society for Peritoneal Dialysis (ISPD) recommendations, "low-risk" peritoneal dialysis (PD)- related peritonitis caused by coagulase-negative staphylococcal species, Streptococcal species, or negative bacterial culture should receive antibiotics for 2 weeks. However, relapsing, recurrent, or repeated episodes are common.

Objectives To compare the incidence of relapsing, recurrent, and repeat peritonitis with a 3-week course, as compared to the conventional 2-week course, antibiotic for PD-related peritonitis. Hypothesis Treatment of low-risk PD-related peritonitis for 3 weeks reduces the incidence of relapsing, recurrent, and repeat peritonitis. Design and subjects Randomized control trial of 310 episodes of "low-risk" PD-related peritonitis.

Study instruments and interventions Patients will be randomized to receive treatment of the effective antibiotic according to the ISPD recommendations for 2 weeks (Conventional Group) or 3 weeks (Extended Group). All patients will be followed for 6 months after completion of treatment. Main outcome measures Complete cure of the peritonitis episode, defined as survival for 6 months without relapsing, recurrent, or repeat peritonitis episodes. Data analysis Data will be analyzed by both intention-to-treat and per protocol approach. The incidences of complete cure, relapsing, recurrent, and repeated peritonitis episodes will be compared. Expected results Based on our pilot study, we expect to find a significantly lower rate of relapsing, recurrent, and repeated peritonitis episodes in the Extended Group. By proving that "low-risk" peritonitis episodes require 3-week course of antibiotic therapy, our result will change the current recommendation and make treatment for 3 weeks course the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* peritonitis episodes caused by CNSS, Streptococcal species, or negative bacterial culture

Exclusion Criteria:

* relapsing peritonitis episodes
* episodes that do not show a clinical response after 5 days of antibiotic therapy
* patients who have difficulty in adhering to the antibiotic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
complete cure | 6 months
  survival without relapsing, recurrent, or repeat peritonitis episodes

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine & Therapeutics, Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No